CLINICAL TRIAL: NCT02022943
Title: Alzheimer's Prevention Registry
Brief Title: Alzheimer's Prevention Registry: A Program to Accelerate Enrollment Into Studies
Acronym: APR
Status: Recruiting | Type: Observational
Sponsor: Banner Health (Other)
Responsible Party: Principal Investigator, Jessica Langbaum, PhD, Senior Director, Research Strategy, Banner Health
Other Study IDs: APR
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Alzheimer's; prevention
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The Alzheimer's Prevention Registry (www.endALZnow.org) will collect contact and demographic information on individuals. The objective is to provide information the latest news and advances in Alzheimer's prevention research, and to inform enrollees about research studies in their community. Enrolled individuals will receive regular email communications. As research studies become available, individuals will be notified via email with information as to how proceed should they be interested. Registry enrollees are under no obligation to participate in a research study. Study opportunities may include surveys, healthy lifestyle interventions (e.g., diet, exercise), memory & thinking tests, brain scans, and investigational drug trials. To join the Registry, please visit www.endALZnow.org

ELIGIBILITY:
Inclusion Criteria:

* Must be able to accept the Alzheimer's Prevention Registry website terms and conditions

Exclusion Criteria:

* None

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anyone who meets entry criteria is eligible to join the Registry.
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2012-05; Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Number of individuals enrolled into Alzheimer's prevention studies | 16 years

SECONDARY OUTCOMES:
Number of individuals referred to Alzheimer's prevention research studies / sites | 16 years

OTHER OUTCOMES:
Total number enrolled into the Alzheimer's Prevention Registry | 16 years

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Langbaum, PhD, Principal Investigator — Banner Alzheimer's Institute
Locations (1):
- Banner Alzheimer's Institute, Phoenix, Arizona, United States

REFERENCES:
- [Result] Langbaum JB, High N, Nichols J, Kettenhoven C, Reiman EM, Tariot PN. The Alzheimer's Prevention Registry: A Large Internet-Based Participant Recruitment Registry to Accelerate Referrals to Alzheimer's-Focused Studies. J Prev Alzheimers Dis. 2020;7(4):242-250. doi: 10.14283/jpad.2020.31. PMID 32920626
- See also: Alzheimer's Prevention Registry — http://www.endALZnow.org